CLINICAL TRIAL: NCT03288246
Title: Point-of-care Viral Load Testing Among HIV-infected Adolescents in Haiti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1708018474
Record Dates: First submitted 2017-09-13; First posted 2017-09-20 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: HIV
Keywords: adolescent; HIV; point-of-care; viral load

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care (No Intervention): Participants in the standard-of-care arm will receive a standard laboratory-based viral load test at baseline, 3, and 6 months.
- Point-of-care (Experimental): Participants in the point-of-care arm will receive a point-of-care viral load test at baseline, 3, and 6 months.
  Interventions: Diagnostic Test: point-of-care viral load test

INTERVENTIONS:
Diagnostic Test: point-of-care viral load test — A point-of-care viral load test returns viral load test results within 90 minutes.
  Arms: Point-of-care

SUMMARY:
This study is designed as an individual randomized trial among 150 HIV-infected adolescents aged 10-24 years who have been on ART for >6 months and will be randomized in a 1:1 fashion to one of two arms: 1) the intervention arm (POC) will receive a POC VL test with adherence counseling informed by the VL result the same day as testing vs. 2) the standard-of-care arm (SOC) will receive a standard laboratory-based test with adherence counseling informed by the VL result 1 month later. The study tests an intervention, POC VL testing, which reduces the time between sample collection and participant receipt of results, thus decreasing the number of steps in the HIV treatment cascade. This intervention was developed to addresses health systems-based barriers which delay clinic, laboratory, and data management processes for VL monitoring for HIV-infected adolescents. Our results will contribute to research on whether POC VL testing is a feasible testing method which could be incorporated into health systems in similar resource-limited settings and whether it can improve outcomes among HIV-infected adolescents.

DETAILED DESCRIPTION:
This study is designed as an individual randomized trial among 150 HIV-infected adolescents aged 10-24 years who have been on ART for >6 months and will be randomized in a 1:1 fashion to one of two arms: 1) the intervention arm (POC) - receiving a POC VL test with adherence counseling informed by the VL result the same day as testing vs. 2) the standard-of-care arm (SOC) - receiving a standard laboratory-based test with adherence counseling informed by the VL result 1 month later. The study tests an intervention, POC VL testing, which reduces the time between sample collection and participant receipt of results, thus decreasing the number of steps in the HIV treatment cascade. This intervention was developed to addresses health systems-based barriers which delay clinic, laboratory, and data management processes for VL monitoring for HIV-infected adolescents. The results will contribute to research on whether POC VL testing is a feasible testing method which could be incorporated into health systems in similar resource-limited settings and whether it can improve outcomes among HIV-infected adolescents. The two study arms are described below.

Standard-of-care (SOC): At the first visit after enrollment and randomization, participants in the SOC arm receive a standard laboratory-based VL test. Steps in the standard laboratory-based VL testing process include: sample collection at a phlebotomy clinic adjacent to the adolescent HIV clinic, labeling and daily storage, transportation (1 hr drive) to the central laboratory, arrival and intake at the laboratory, processing in the fully automated Abbott system, manual entry of the printed results into an excel spreadsheet by laboratory staff, and manual entry of results on the spreadsheet into the EMR by data management staff. This process - from sample collection to patient return of results - varies depending on the volume of samples collected each day and on laboratory and data management staffing. Average time from blood collection to availability of the result in the EMR is 2-3 weeks. Per standard clinical care at the adolescent HIV clinic, adolescents return for monthly visits, and the patient receives the VL result and adherence counseling which is informed by the VL result 1 month after providing the blood sample. The primary endpoint is return of the VL result within 6 weeks of sample collection to allow for a short time buffer for appointments that are not scheduled exactly 1 month from the previous visit for reasons related to school, work, family obligations, or holidays.

These standard laboratory procedures were developed to meet the high demand for VL testing when the Haitian national guidelines switched from recommending routine CD4 testing to routine VL testing. Since the Abbott systems are fully automated and can batch large quantities of samples together, this approach is appropriate for a routine nation-wide health system testing protocol. However, the need for transportation, cold-chain storage, and manual entry of thousands of results every year may not be the optimal structure for HIV-infected adolescents who are more likely to have high VL results and are more likely to be lost from care in between visits. This study will test the POC VL test vs. this standard laboratory-based test to determine if reducing the time between sample collection and patient receipt of results (removing a step in the HIV treatment cascade), can increase the impact of VL testing on clinical management and adolescent patient outcomes. The study will test if implementation of the POC VL test, in collaboration with clinicians and laboratory staff, and accompanied by patient education, can address many of the logistical barriers to laboratory-based VL testing in a resource-limited setting such as Haiti.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10-24 years
* HIV-infected
* On ART for > 6 months
* Permanent residence in Port-au-Prince
* Able to provide informed consent/assent

Exclusion Criteria:

* Requires urgent VL test the day of enrollment/randomization
* Requires ART regimen change
* Currently pregnant
* Co-infected with tuberculosis
* Severe co-morbidities including cognitive impairment, bipolar disorder, psychosis, or current need for inpatient psychiatric hospitalization

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
The number of steps in the HIV care cascade involved with viral load testing. | 1 day of clinic visit
  The number of steps within the HIV care cascade involved with viral load testing will be measured comparing standard laboratory-based testing to POC testing.

SECONDARY OUTCOMES:
The proportion of participants who demonstrate comprehension of the correlation between ART adherence and viral level | 1 month
  The proportion of participants who demonstrate comprehension of the correlation between ART adherence and viral level 1 month after receiving their VL test result will be measured.
The proportion of participants who achieve or sustain a viral level <1000 cells/ml | 6 months
  The proportion of participants who achieve or sustain a viral level <1000 cells/ml 6 months from the index VL test will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fitzgerald, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- GHESKIO, Port-au-Prince, Haiti

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared once the trial is complete

REFERENCES:
- [Derived] Reif LK, Belizaire ME, Rouzier V, Seo G, Severe P, Bajo Joseph JM, Joseph B, Apollon S, Pape JW, McNairy ML, Elul B, Fitzgerald DW, Arpadi SM, Abrams EJ, Kuhn L. Point-of-care viral load testing among adolescents and young adults living with HIV in Haiti: a randomized control trial. AIDS Care. 2022 Apr;34(4):409-420. doi: 10.1080/09540121.2021.1981816. Epub 2021 Oct 6. PMID 34612092
- [Derived] Reif LK, Belizaire ME, Seo G, Rouzier V, Severe P, Joseph JM, Joseph B, Apollon S, Abrams EJ, Arpadi SM, Elul B, Pape JW, McNairy ML, Fitzgerald DW, Kuhn L. Point-of-care viral load testing among adolescents and youth living with HIV in Haiti: a protocol for a randomised trial to evaluate implementation and effect. BMJ Open. 2020 Aug 31;10(8):e036147. doi: 10.1136/bmjopen-2019-036147. PMID 32868354